CLINICAL TRIAL: NCT05025423
Title: Phase II Trial of Venetoclax and Rituximab as Initial Therapy in Older Patients With Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study sponsor withdrew funding early, forcing this study to stop all activity and close pre-maturely.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J2146; IRB00288478 (Other: JHM IRB)
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — venetoclax; Rituximab

STUDY DESIGN:
Intervention Model Description: Venetoclax dose escalation for Cycles 1-4. If Complete response (CR) at Cycle 4, continue with cycles 5-12 at fixed venetoclax 400mg dose. If partial response (PR) at Cycle 4, continue with cycles 5-8 at fixed venetoclax 800mg dose. If CR at Cycle 8 after PR, continue with cycles 9-12 at fixed venetoclax 800mg dose. If continued PR at Cycle 8, reduce venetoclax to 400mg and add bendamustine 90 mg/m2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- venetoclax and rituximab in patients over 60 yrs old with previously untreated mantle cell lymphoma (Experimental): Venetoclax dose escalation for Cycles 1-4. If Complete response (CR) at Cycle 4, continue with cycles 5-12 at fixed venetoclax 400mg dose. If partial response (PR) at Cycle 4, continue with cycles 5-8 at fixed venetoclax 800mg dose. If CR at Cycle 8 after PR, continue with cycles 9-12 at fixed venetoclax 800mg dose. If continued PR at Cycle 8, reduce venetoclax to 400mg and add bendamustine 90 mg/m2.
  Interventions: Drug: Venetoclax Oral Tablet [Venclexta]

INTERVENTIONS:
Drug: Venetoclax Oral Tablet [Venclexta] — Sequential dose levels for Venetoclax dependent on patient response. Fixed doses of 375 mg/m2 rituximab. Fixed dose of Bendamustine 90 mg/m2 added for those with continued PR at Cycle 8
  Other Names: rituximab infusion [Rituxan]; Bendamustine infusion

SUMMARY:
The proposed study is an open-label, single arm phase II study of venetoclax in combination with rituximab in patients over the age of 60 with previously untreated mantle cell lymphoma. The primary objective of the trial is to determine whether the combination of venetoclax with rituximab in this patient population yields a clinically acceptable proportion of overall responses (ORR, assessed by PET/CT with Lugano criteria) without chemotherapy.

DETAILED DESCRIPTION:
For young, fit patients with mantle cell lymphoma, intensive chemotherapy and rituximab followed by ASCT is often used to achieve prolonged disease free survival. However, this therapy is not curative and has not been shown to improve overall survival. For older or frail patients, who are ineligible for stem cell transplantation, improved disease free survival can be achieved with chemotherapy and rituximab without ASCT, but at the cost of significant short and long-term toxicity. Venetoclax monotherapy has shown impressive single-agent activity in relapsed and refractory mantle cell lymphoma with low rates of adverse events.

The hypothesis is that initial therapy with venetoclax and rituximab will result in rates of CR and PR that are comparable to historical rates with chemoimmunotherapy. Furthermore, this regimen will have fewer side effects than traditional therapy. Investigators also hypothesize that patients achieving a CR will have long durations of response that will continue after stopping venetoclax.

Study investigators will test this hypothesis with an open label, single arm phase II trial with a target accrual of 40 participants. This study will include patients over age 60 who are not candidates for aggressive upfront therapy . Subjects will receive venetoclax and rituximab for up to 12 cycles of 4 weeks each. All patients will stop venetoclax after 12 cycles. Participants who have stable disease or disease progression after 4 cycles will be removed from the trial in order to receive standard of care chemoimmunotherapy. Participants who do not achieve a CR after 8 cycles of venetoclax and rituximab will receive 4 cycles of standard of care bendamustine in addition to continuing rituximab and venetoclax.

This is the first phase II study of venetoclax and rituximab alone as initial therapy for mantle cell lymphoma. In the relapsed and refractory setting, venetoclax has shown high activity in MCL, and as such is a promising option for a non-chemotherapy approach to upfront treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically confirmed diagnosis of mantle cell lymphoma as defined by the World Health Organization (WHO) classification scheme.
* Age ≥ 60
* Subjects must be previously untreated for mantle cell lymphoma and deemed to require treatment by the treating physician
* ECOG performance status of 0-3
* Subject must have adequate bone marrow* without growth factor support as follows:

  * Absolute Neutrophil Count (ANC) ≥ 1000/μL
  * Platelets ≥ 75,000/mm3 (entry platelet count must be independent of transfusion within 14 days of Screening)
  * Hemoglobin ≥ 9.0 g/dL * These criteria may be waived by study investigators if there is evidence of bone marrow involvement by MCL that is believed to be the cause of the cytopenias.
* Subject must have adequate renal, and hepatic function, per laboratory reference range at screening as follows:

  * Subject must have adequate renal, and hepatic function, per laboratory reference range at screening as follows:
  * Calculated creatinine clearance ≥ 40 mL/min; determined via the Cockcroft-Gault formula.
  * AST and ALT ≤ 3.0 × ULN; Bilirubin ≤ 1.5 × ULN*. Subjects with Gilbert's Syndrome may have a bilirubin > 1.5 × ULN

    * These criteria may be waived by study investigators if abnormal values believed to be due to lymphoma.
* Female subjects must be surgically sterile, postmenopausal (for at least 1 year), or have negative results for a pregnancy test performed as follows:

  * At Screening on a serum sample obtained within 14 days prior to the first study drug administration, and
  * Prior to dosing on a urine sample obtained on Cycle 1 Day 1 if it has been > 7 days since obtaining the serum pregnancy test results.
  * All female subjects not surgically sterile or postmenopausal (for at least 1 year) and non-vasectomized male subjects must practice at least 1 of the following methods of birth control:

    1. Total abstinence from sexual intercourse (minimum 1 complete menstrual cycle);
    2. A vasectomized partner(s);
    3. Hormonal contraceptives (oral, parenteral, vaginal ring or transdermal) for at least 3 months prior to study drug administration;
    4. Double-barrier method (condoms and diaphragm with spermicidal [sponge, jellies or creams]).
* Ability to understand and willingness to sign IRB-approved informed consent

Exclusion Criteria:

* Subject has blastoid-variant mantle cell lymphoma
* Subject requires immediate cytoreduction as determined by study investigators
* Subject has documented CNS involvement of mantle cell lymphoma
* Subject has Ann Arbor stage I or contiguous stage II mantle cell lymphoma
* Subject has an uncontrolled infection
* Subject has HIV infection
* All subjects will be screened for Hepatitis B (HBsAg, anti-HBs, anti-HBc IgM and total) and Hepatitis C (antibody or RNA). Subjects who are positive for Hepatitis B by HBsAg or DNA as well as subjects positive for Hepatitis C will be excluded. Subjects with anti-HBc positivity and DNA negative may be included but will be required to undergo monthly HBV DNA testing and liver function liver function testing (AST, ALT, alkaline phosphatase, total bilirubin). Patients with HCV antibody positivity and HCV pcr negativity are eligible to be included.
* Subject requires the use of warfarin
* Subject has received immunization with live virus vaccine within 28 days prior to the first dose of study drug
* A female subject is pregnant or breast-feeding

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) after four cycles of venetoclax and rituximab. | 120 days
  The ORR will be the sum of complete (CR) and partial responses (PR)as determined by PET/CT and Lugano criteria. Simon's optimal two-stage design will be used to test the null hypothesis that the true ORR is 50% or less (not considered clinically acceptable).

SECONDARY OUTCOMES:
Proportion of CR | 120 days
  Proportion of CR as determined by PET/CT and Lugano criteria after four cycles
Proportion of PR | 120 days
  Proportion of PR as determined by PET/CT and Lugano criteria after four cycles
Proportion of stable disease | 120 days
  Proportion of stable disease as determined by PET/CT and Lugano criteria after four cycles
Proportion of disease progression | 120 days
  Proportion of disease progression as determined by PET/CT and Lugano criteria after four cycles
Rate of CR after 8 cycles of venetoclax and rituximab | 240 days
  Rate of CR as determined by PET/CT and Lugano criteria after 8 cycles of venetoclax and rituximab
Rate of PR after 8 cycles of venetoclax and rituximab | 240 days
  Rate of PR as determined by PET/CT and Lugano criteria after 8 cycles of venetoclax and rituximab
Proportion of progression free survival (PFS) | 240 days
  To evaluate the progression free survival (PFS) in the intent to treat (ITT) population
free survival (PFS) | 240 days
  To evaluate the progression free survival (PFS) in the intent to treat (ITT) population
overall survival (OS) | 240 days
  To evaluate the overall survival (OS) in the intent to treat (ITT) population
duration of response (DOR) | 240 days
  To evaluate the duration of response (DOR) for participants achieving a CR or PR

CONTACTS AND LOCATIONS:
Overall Officials: Lode Swinnen, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States